CLINICAL TRIAL: NCT05621460
Title: The Effect of Water Carbonation on Orthostatic Tolerance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Simon Fraser University (Other)
Responsible Party: Principal Investigator, Dr. Victoria Claydon, Professor, Simon Fraser University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 30000955
Record Dates: First submitted 2022-11-10; First posted 2022-11-18 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Orthostatic Hypotension; Syncope; Vasovagal Syncope
Keywords: Tilt table; Osmopressor reflex; Gastropressor reflex
MeSH Terms: conditions — Hypotension, Orthostatic; Syncope; Syncope, Vasovagal | interventions — Carbonated Water

STUDY DESIGN:
Intervention Model Description: Each participant will complete the test for every condition (3 tests per participant, order of treatment randomized).
Who Masked: Investigator
Masking Description: The investigator determining the end of the test (the time to presyncope) will be blinded to the condition.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 500mL carbonated water first, then 500mL of still water, then 50mL of still water (Experimental): Participants will undergo this test on three separate days. On each day participants will be asked to drink a glass of water: either a 50mL drink of still water (control condition), a 500mL drink of still (non-carbonated) water, or a 500mL drink of carbonated water. In this arm of the study, participants will receive 500mL carbonated water on the first test day, 500mL still water on the second test day, then 50mL still water on the third day.
  Interventions: Other: 500mL carbonated water; Other: 500mL still water; Other: 50mL still water
- 500mL still water first, then 500 mL carbonated water, then 50mL still water (Experimental): Participants will undergo this test on three separate days. On each day participants will be asked to drink a glass of water: either a 50mL drink of still water (control condition), a 500mL drink of still (non-carbonated) water, or a 500mL drink of carbonated water. In this arm of the study, participants will receive 500mL still water on the first test day, 500mL carbonated water on the second test day, then 50mL still water on the third day.
  Interventions: Other: 500mL carbonated water; Other: 500mL still water; Other: 50mL still water
- 500mL carbonated water first, then 50mL of still water, then 500mL of still water (Experimental): Participants will undergo this test on three separate days. On each day participants will be asked to drink a glass of water: either a 50mL drink of still water (control condition), a 500mL drink of still (non-carbonated) water, or a 500mL drink of carbonated water. In this arm of the study, participants will receive 500mL carbonated water on the first test day, 50mL still water on the second test day, then 500mL still water on the third day.
  Interventions: Other: 500mL carbonated water; Other: 500mL still water; Other: 50mL still water
- 500mL still water first, then 50mL still water, then 500 mL carbonated water (Experimental): Participants will undergo this test on three separate days. On each day participants will be asked to drink a glass of water: either a 50mL drink of still water (control condition), a 500mL drink of still (non-carbonated) water, or a 500mL drink of carbonated water. In this arm of the study, participants will receive 500mL still water on the first test day, 50mL still water on the second test day, then 500mL carbonated water on the third day.
  Interventions: Other: 500mL carbonated water; Other: 500mL still water; Other: 50mL still water
- 50mL still water first, then 500mL still water, then 500 mL carbonated water (Experimental): Participants will undergo this test on three separate days. On each day participants will be asked to drink a glass of water: either a 50mL drink of still water (control condition), a 500mL drink of still (non-carbonated) water, or a 500mL drink of carbonated water. In this arm of the study, participants will receive 50mL still water on the first test day, 500mL carbonated water on the second test day, then 500mL carbonated water on the third day.
  Interventions: Other: 500mL carbonated water; Other: 500mL still water; Other: 50mL still water
- 50mL still water first, then 500mL carbonated water, then 500 mL still water (Experimental): Participants will undergo this test on three separate days. On each day participants will be asked to drink a glass of water: either a 50mL drink of still water (control condition), a 500mL drink of still (non-carbonated) water, or a 500mL drink of carbonated water. In this arm of the study, participants will receive 50mL still water on the first test day, 500mL still water on the second test day, then 500mL still water on the third day.
  Interventions: Other: 500mL carbonated water; Other: 500mL still water; Other: 50mL still water

INTERVENTIONS:
Other: 500mL carbonated water — Drink 500mL carbonated water immediately prior to head-up tilt test
Other: 500mL still water — Drink 500mL still water immediately prior to head-up tilt test
Other: 50mL still water — Drink 50mL still water immediately prior to head-up tilt test

SUMMARY:
The primary purpose of this investigation is to determine whether water carbonation can improve orthostatic tolerance in healthy control volunteers. Orthostatic tolerance refers to the ability to maintain an adequate blood pressure when standing. In some individuals blood pressure can fall when standing, predisposing to dizzy spells or fainting episodes. Drinking water can boost blood pressure and making fainting episodes less likely. However, it is not clear whether the carbonation of the water has any further impact on the blood pressure response. This is important because it may be that carbonated water expands the stomach (gastric distension), provoking an increase in sympathetic activity. The increase in sympathetic nervous system activity boosts blood pressure. Resolving this question would have important implications for patients with syncope. This study will test whether carbonated water will have any further impact on blood pressure than the already known effect of non-carbonated water.

DETAILED DESCRIPTION:
The primary purpose of this investigation is to determine whether water carbonation can improve orthostatic tolerance in healthy control volunteers. Orthostatic tolerance refers to the ability to maintain an adequate blood pressure when standing [1]. In some individuals blood pressure can fall when standing, predisposing to dizzy spells or fainting episodes [1]. Drinking water can boost blood pressure and making fainting episodes less likely [2-8]. However, it is not clear whether the carbonation of the water has any further impact on the blood pressure response [9,10]. This is important because it may be that carbonated water expands the stomach (gastric distension), provoking an increase in sympathetic activity. The increase in sympathetic nervous system activity boosts blood pressure. Resolving this question would have important implications for patients with syncope. This study will test whether carbonated water will have any further impact on blood pressure than the already known effect of non-carbonated water.

Volunteers (n=25) will be asked to undergo a "tilt test" to assess cardiovascular reflex control and orthostatic tolerance (measured as time to presyncope, or near fainting, in minutes). It has been previously shown that this technique to be reproducible, reliable, and to have high sensitivity and specificity for differentiating persons with differing orthostatic tolerance, or for examining the effects of interventions aimed at improving orthostatic tolerance [4,6,11-18].

Volunteers will undergo this test on three separate days. On each day participants will be asked to drink a glass of water: either a 50ml drink of room temperature water (control condition), a 500ml drink of flat (non-carbonated) room temperature water, or a 500ml drink of carbonated room temperature water. The study will be conducted in a randomised, single-blind fashion. The investigator responsible for terminating the test will be blinded as to the water condition on each test day, rendering the study single blind. It will not be possible to blind participants as to the carbonation of the water, however, participants will not be informed as to the hypothesised impact of the water conditions.

ELIGIBILITY:
Inclusion Criteria:

* healthy, English-speaking

Exclusion Criteria:

* pregnancy or suspected pregnancy, history of cardiovascular disease, history of neurological disease, history of recurrent fainting (≥ 2 episodes of fainting with loss of consciousness in the prior 6 months)

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Orthostatic tolerance | 0-50 minutes
  The time, in minutes, to presyncope (near-fainting) after the initiation of head-up tilt

CONTACTS AND LOCATIONS:
Overall Officials: Victoria E Claydon, PhD, Principal Investigator — Professor, Biomedical Physiology and Kinesiology
Locations (1):
- Simon Fraser University, Burnaby, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
Data will be presented in aggregate form and no identifiers will be included.

REFERENCES:
- [Background] Hainsworth R, Claydon V E. Syncope and fainting: classification and physiological basis. In: Bannister R, Mathias CJ, eds. Autonomic failure: a textbook of clinical disorders of the autonomic nervous system. Oxford: Oxford University Press, 2006
- [Background] Mathias CJ. A 21st century water cure. Lancet. 2000 Sep 23;356(9235):1046-8. doi: 10.1016/S0140-6736(00)02723-9. PMID 11009136
- [Background] Mathias CJ, Young TM. Water drinking in the management of orthostatic intolerance due to orthostatic hypotension, vasovagal syncope and the postural tachycardia syndrome. Eur J Neurol. 2004 Sep;11(9):613-9. doi: 10.1111/j.1468-1331.2004.00840.x. PMID 15379740
- [Background] Schroeder C, Bush VE, Norcliffe LJ, Luft FC, Tank J, Jordan J, Hainsworth R. Water drinking acutely improves orthostatic tolerance in healthy subjects. Circulation. 2002 Nov 26;106(22):2806-11. doi: 10.1161/01.cir.0000038921.64575.d0. PMID 12451007
- [Background] Brown CM, Barberini L, Dulloo AG, Montani JP. Cardiovascular responses to water drinking: does osmolality play a role? Am J Physiol Regul Integr Comp Physiol. 2005 Dec;289(6):R1687-92. doi: 10.1152/ajpregu.00205.2005. Epub 2005 Jul 21. PMID 16037127
- [Background] Claydon VE, Schroeder C, Norcliffe LJ, Jordan J, Hainsworth R. Water drinking improves orthostatic tolerance in patients with posturally related syncope. Clin Sci (Lond). 2006 Mar;110(3):343-52. doi: 10.1042/CS20050279. PMID 16321141
- [Background] Lu CC, Diedrich A, Tung CS, Paranjape SY, Harris PA, Byrne DW, Jordan J, Robertson D. Water ingestion as prophylaxis against syncope. Circulation. 2003 Nov 25;108(21):2660-5. doi: 10.1161/01.CIR.0000101966.24899.CB. Epub 2003 Nov 17. PMID 14623807
- [Background] Boschmann M, Steiniger J, Hille U, Tank J, Adams F, Sharma AM, Klaus S, Luft FC, Jordan J. Water-induced thermogenesis. J Clin Endocrinol Metab. 2003 Dec;88(12):6015-9. doi: 10.1210/jc.2003-030780. PMID 14671205
- [Background] May M, Jordan J. The osmopressor response to water drinking. Am J Physiol Regul Integr Comp Physiol. 2011 Jan;300(1):R40-6. doi: 10.1152/ajpregu.00544.2010. Epub 2010 Nov 3. PMID 21048076
- [Background] Jordan J, Shannon JR, Black BK, Ali Y, Farley M, Costa F, Diedrich A, Robertson RM, Biaggioni I, Robertson D. The pressor response to water drinking in humans : a sympathetic reflex? Circulation. 2000 Feb 8;101(5):504-9. doi: 10.1161/01.cir.101.5.504. PMID 10662747
- [Background] Al Shamma YMA, Hainsworth R. A quantitative comparison of the circulatory responses in humans to graded upright tilting and graded lower body negative pressure. Cardiogenic Reflexes (1987):431-432.
- [Background] Brown CM, Hainsworth R. Forearm vascular responses during orthostatic stress in control subjects and patients with posturally related syncope. Clin Auton Res. 2000 Apr;10(2):57-61. doi: 10.1007/BF02279892. PMID 10823336
- [Background] Bush VE, Wight VL, Brown CM, Hainsworth R. Vascular responses to orthostatic stress in patients with postural tachycardia syndrome (POTS), in patients with low orthostatic tolerance, and in asymptomatic controls. Clin Auton Res. 2000 Oct;10(5):279-84. doi: 10.1007/BF02281110. PMID 11198483
- [Background] Claydon VE, Hainsworth R. Salt supplementation improves orthostatic cerebral and peripheral vascular control in patients with syncope. Hypertension. 2004 Apr;43(4):809-13. doi: 10.1161/01.HYP.0000122269.05049.e7. Epub 2004 Feb 23. PMID 14981050
- [Background] Claydon VE, Hainsworth R. Cerebral autoregulation during orthostatic stress in healthy controls and in patients with posturally related syncope. Clin Auton Res. 2003 Oct;13(5):321-9. doi: 10.1007/s10286-003-0120-8. PMID 14564654
- [Background] el-Bedawi KM, Hainsworth R. Combined head-up tilt and lower body suction: a test of orthostatic tolerance. Clin Auton Res. 1994 Apr;4(1-2):41-7. doi: 10.1007/BF01828837. PMID 8054836
- [Background] Cooper VL, Hainsworth R. Carotid baroreceptor reflexes in humans during orthostatic stress. Exp Physiol. 2001 Sep;86(5):677-81. doi: 10.1113/eph8602213. PMID 11571497
- [Background] Cooper VL, Hainsworth R. Effects of dietary salt on orthostatic tolerance, blood pressure and baroreceptor sensitivity in patients with syncope. Clin Auton Res. 2002 Aug;12(4):236-41. doi: 10.1007/s10286-002-0018-x. PMID 12357276